CLINICAL TRIAL: NCT06082648
Title: Observation and Intervention Study of Brain-Gut Function Reconstruction After Intersphincteric Resection (ISR) for Ultra-Low Rectal Tumors
Brief Title: Study of Brain-Gut Function Reconstruction After Intersphincteric Resection for Ultra-Low Rectal Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jianbin Xiang, Professor，Ph.D., M.D., Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2023-087
Record Dates: First submitted 2023-09-27; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Rectal Neoplasms
Keywords: Ultra-low rectal tumors; Intersphincteric Resection; transcranial magnetic stimulation; fMRI
MeSH Terms: conditions — Rectal Neoplasms | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Stimultion Group (Sham Comparator): Patients on the Sham stimulation group will be interfered with the stimulation coil perpendicular to the skull, so that they will hear the sound of machine without having therapeutic effects. The parameters will be the same as those in the stimulation group.
  Interventions: Device: Sham Transcranial magnetic stimulationt
- Pre-ileostomy-closure Stimultion Group (Active Comparator): Patients on the Pre-ileostomy-closure group will be interfered with stimulation 3 weeks before the procedure of ileostomy closure.
  Interventions: Device: Transcranial magnetic stimulation
- Post-ileostomy-closure Stimultion Group (Active Comparator): Patients on the Post-ileostomy-closure group will be interfered with stimulation 3 weeks after the procedure of ileostomy closure.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — The magnetic stimulator equipment is provided by the MagProX100 magnetic stimulator ( MagVenture, Lucernemarken, DK-3520 Farum, Denmark), with 8-shaped coil, a maximum stimulation frequency of 30Hz and a maximum stimulation intensity of 6 Tesla.Stimulation group: Intermittentpulse transcranial magnetic stimulation (iTBS) will be performed with : the cluster consists of 3 pulses, the intra-cluster frequency is 50Hz, the intercluster frequency is 5Hz, the interval is 8.2s for every stimulus. There are 20 cycles and a total of 600 pulses. Each intervention time is 3min11s, and the stimulation intensity is set as 80% resting state motion threshold. The intervention will be performed once a day for 2 weeks.
  Arms: Post-ileostomy-closure Stimultion Group; Pre-ileostomy-closure Stimultion Group
Device: Sham Transcranial magnetic stimulationt — The magnetic stimulator equipment is provided by the MagProX100 magnetic stimulator ( MagVenture, Lucernemarken, DK-3520 Farum, Denmark), with 8-shaped coil, a maximum stimulation frequency of 30Hz and a maximum stimulation intensity of 6 Tesla. Patients on the Sham stimulation group will be interfered with the stimulation coil perpendicular to the skull, so that they will hear the sound of machine without having therapeutic effects. The parameters will be the same as those in the stimulation group.
  Arms: Sham Stimultion Group

SUMMARY:
To investigate the effects of intersphincteric resection (ISR) of ultra-low rectal tumor on the brain-rectoanal function of patients, and to precisely localize the cerebral functional regulatory regions for intervention targets of anorectal remodeling. Utilizing transcranial magnetic stimulation(TMS) technology to explore the functional remodeling of the "new" anorectal muscle groups and provide a theoretical basis for more research on the rehabilitation and mechanism of fecal incontinence.

DETAILED DESCRIPTION:
This study is a Single-center Phase II, Open, Three-Arm clinical trial. We prospectively enroll patients who undergo ISR for ultra-low rectal tumor in the department of General Surgery, Huashan Hospital, Fudan University. Patients with ileostomy closure are randomly divided into two groups (TMS group and false stimulation group), and healthy volunteers were recruited. The differences of task-state fMRI between healthy volunteers, and ISR patients (both preoperative and postoperative) are compared, combined with rectal function scores (Wexner score, LARS score) and quality of life scale (EORTC QLQ-C30, EORTC QLQ-CR38). Proctoanal manometry are used to find the precise location of the proctoanal motor function area in the cerebral cortex, and to evaluate the effect and value of TMS on postoperative anorectal motor function remodeling in patients with ISR.

ELIGIBILITY:
Inclusion Criteria:

* Primary ultra-low rectal tumor patient who is received intersphincteric resection and preventive ileostomy was performed.
* Patient who is willing to participate in the study, and voluntarily sign informed consent.

Exclusion Criteria:

* Anastomotic leakage or other serious complications occur after surgery.
* Advanced tumor, tumor recurrence or metastasis.
* Patients with contraindications of fMRI scanning, such as history of metal implants in the body, claustrophobia, etc.
* Patients with contraindications for TMS treatment, such as intracranial metal implants, epilepsy history, heart disease with unstable heart function, retinal detachment, etc.
* Combined with organic brain disease and drug abuse history.
* Combined with other mental diseases.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
The differences of cortical activated areas in task-state fMRI in ISR patients. | pre-ISR, pre-ileostomy closure, 6,12 month after ileostomy closure.
  Cortical activated areas in BOLD sequence of patients in different time frame
The differences of cortical activated areas in task-state fMRI between health volunteers and postoperative ISR patients. | 12 month after ileostomy closure。
  Cortical activated areas in BOLD sequence of health volunteers and patients
Rectal function scores (Wexner score) | pre-ISR，1, 3 , 6, 9, 12, 18, 24 month after ileostomy closure.
  Wexner score of patients in different time frame
Rectal function scores (LARS score) | pre-ISR，1, 3 , 6, 9, 12, 18, 24 month after ileostomy closure.
  LARS score of patients in different time frame
Quality of life Scale (EORTC QLQ-C30) | pre-ISR，1, 3 , 6, 9, 12, 18, 24 month after ileostomy closure.
  EORTC QLQ-C30 of patients in different time frame
Quality of life Scale (EORTC QLQ-CR38) | pre-ISR，1, 3 , 6, 9, 12, 18, 24 month after ileostomy closure.
  EORTC QLQ-CR38 of patients in different time frame

SECONDARY OUTCOMES:
Proctoanal manometry | pre-ISR，3 , 6, 12, 18, 24 month after ileostomy closure.
  Proctoanal manometry of Patients in different time frame

CONTACTS AND LOCATIONS:
Overall Officials: Jianbin Xiang, PhD, Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China